CLINICAL TRIAL: NCT00997386
Title: A Phase II Study of Reduced-Intensity Allogeneic Peripheral Blood Stem Cell Transplantation (PBSCT) for Treatment of Hematologic Malignancies and Hematopoietic Failure States
Brief Title: Reduced Intensity Allogeneic PBSCT to Treat Hematologic Malignancies and Hematopoietic Failure States
Acronym: ALBUM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-0679-04
Record Dates: First submitted 2009-10-15; First posted 2009-10-19 (Estimated); Results first posted 2018-12-24 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Hematologic Neoplasms; Multiple Myeloma; Anemia, Aplastic; Hemoglobinuria, Paroxysmal; Myelofibrosis
Keywords: Hematologic malignancies; lymphoma, leukemia, MDS (myelodysplastic syndrome); reduced-intensity preparative regimen; allogeneic peripheral blood stem cell transplant; myelofibrosis or other myeloproliferative syndromes
MeSH Terms: conditions — Hematologic Neoplasms; Multiple Myeloma; Anemia, Aplastic; Hemoglobinuria, Paroxysmal; Primary Myelofibrosis; Lymphoma; Leukemia; Myelodysplastic Syndromes | interventions — Busulfan; Melphalan; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- busulfan, and melphalan, and alemtuzumab (Experimental): Three drug regimen using busulfan, and melphalan, and alemtuzumab.
  Interventions: Drug: busulfan, and melphalan, and alemtuzumab

INTERVENTIONS:
Drug: busulfan, and melphalan, and alemtuzumab — intravenous busulfan 3.2 mg/kg/dose daily for 2 days, on days -5 and -4 (i.e., 5 and 4 days, respectively, before PBSCT).
  intravenous melphalan 100 mg/m2 on day -3.
  intravenous alemtuzumab 30 mg/dose for 2 days, on days -2 and -1.
  Other Names: Busulfan (Busulfex®),; Melphalan (Alkeran®); Alemtuzumab (Campath®)

SUMMARY:
The purpose of this study is to look at whether the combination of lower-dose chemotherapy with two chemotherapy (anti-cancer) drugs, called busulfan and melphalan, and an antibody medication called alemtuzumab (Campath®), can prevent rejection of donor blood stem cells so that those cells take hold and build a healthy new blood cell factory after transplant. The study will also look at the safety of the combination of drugs and of the transplant of peripheral blood stem cells from a healthy relative or an unrelated donor.

DETAILED DESCRIPTION:
Transplantation of related or unrelated allogeneic peripheral blood stem cells (PBSCs) after administration of a reduced-intensity regimen of busulfan, melphalan and alemtuzumab will be associated with satisfactory engraftment and acceptable post-transplant non-relapse mortality.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 to 75 years or age 18 to 49 with one or more of these risk factors: prior autologous, allogeneic or syngeneic HCT (Hematopoietic cell transplantation); not in first complete remission or first chronic phase; and/or presence of one or more medical conditions that would place the subject at high risk such as heart and kidney disease.
* Subjects with hematologic cancers must have received at least one previous course of chemotherapy or biological therapy. In other words, the subject cannot enroll in this trial for initial treatment of the disease.
* Availability of a healthy related or unrelated volunteer allogeneic donor.

Exclusion Criteria:

* Eligible for another study or standard of care treatment that offers higher probability of cure or long-term control of subject's disease.
* Severe abnormal function of organs such as heart, kidneys, liver.
* Untreated or progressive central nervous system involvement by the disease.
* Subject is pregnant or breast-feeding.
* Performance score is below 50: at the least, requires considerable assistance and frequent medical care.
* Positive for the HIV [AIDS] virus
* Life expectancy less than 12 weeks with conventional treatments.
* For subjects capable of having children, refusal to practice birth control while on this study and for at least 12 months after PBSCT or after stopping post-transplant immunosuppressive treatments, whichever occurs later.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-09; Primary Completion 2014-04 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew M Yeager, MD, Principal Investigator — University of Arizona
Locations (1):
- University Medical Center and UMC-North Clinic, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Busulfan, and Melphalan, and Alemtuzumab: Three drug regimen using busulfan, and melphalan, and alemtuzumab.
  Busulfan, and melphalan, and alemtuzumab: intravenous busulfan 3.2 mg/kg/dose daily for 2 days, on days -5 and -4 (i.e., 5 and 4 days, respectively, before PBSCT).
  Intravenous melphalan 100 mg/m2 on day -3.
  Intravenous alemtuzumab 30 mg/dose for 2 days, on days -2 and -1.
Period: Overall Study
Arm/Group | Busulfan, and Melphalan, and Alemtuzumab
Started | 16
Completed | 9
Not Completed | 7
Not completed — Death | 7

BASELINE CHARACTERISTICS:
Arm/Group | Busulfan, and Melphalan, and Alemtuzumab
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Presence of Donor Lymphohematopoietic Chimerism (Defined as at Least 50% Donor Cells in the Peripheral Blood) in Peripheral Blood by Day +100 (i.e., 100 Days After Allogeneic PBSCT).
Description: To determine the efficacy of related or unrelated allogeneic PBSC transplantation (PBSCT) using a preparative regimen of busulfan, melphalan and alemtuzumab, as measured by durable donor lymphohematopoietic cell engraftment. The primary efficacy endpoint is the presence of donor lymphohematopoietic chimerism (defined as at least 50% donor cells in the peripheral blood) in peripheral blood by day +100 (i.e., 100 days after allogeneic PBSCT).
Time Frame: Day +100
Population: Data were collected but could not be analyzed. PI for this study has retired and any data that were gathered, are lost. No data are available for this assessment
Arm/Group | Busulfan, and Melphalan, and Alemtuzumab
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Relapse-free Survival.
Description: To determine the safety of related or unrelated allogeneic PBSCT using a preparative regimen of busulfan, melphalan and alemtuzumab. The primary safety endpoint is non-relapse mortality at day +100.
Time Frame: Day +100
Population: as for outcome 1
Arm/Group | Busulfan, and Melphalan, and Alemtuzumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Event-free Survival.
Description: as for outcome 2
Time Frame: Day +100
Population: as for outcome 1
Arm/Group | Busulfan, and Melphalan, and Alemtuzumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Number of Participants With Overall Survival.
Description: as for outcome 2
Time Frame: Day +100
Population: as for outcome 1
Arm/Group | Busulfan, and Melphalan, and Alemtuzumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Busulfan, and Melphalan, and Alemtuzumab
All-Cause Mortality (participants affected / at risk) | 7/16
Serious Adverse Events (participants affected / at risk) | 3/16
Other Adverse Events (participants affected / at risk) | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Busulfan, and Melphalan, and Alemtuzumab (N=16)
Pneumatosis cystoides intestinalis (Gastrointestinal disorders) | 1
Fever (General disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Busulfan, and Melphalan, and Alemtuzumab (N=16)
Respiratory Acidosis (Respiratory, thoracic and mediastinal disorders) | 1
Adult Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Hypoalbuminemia (Blood and lymphatic system disorders) | 2
Alkaline phosphatase (Blood and lymphatic system disorders) | 2
Respiratory Alkalosis (Respiratory, thoracic and mediastinal disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Anorexia (Metabolism and nutrition disorders) | 4
Hyperbilirubinemia (Blood and lymphatic system disorders) | 2
Bladder spasms (Renal and urinary disorders) | 1
Blood/Bone marrow - other (Blood and lymphatic system disorders) | 5
Hypocalcemia (Blood and lymphatic system disorders) | 1
Cardiac arrhythmia (Cardiac disorders) | 2
Cardiac - general (Cardiac disorders) | 3
Infectious colitis (Gastrointestinal disorders) | 1
Confusion (General disorders) | 2
Constipation (Gastrointestinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Creatinine (Blood and lymphatic system disorders) | 10
Skin - other (Skin and subcutaneous tissue disorders) | 6
Diarrhea (Gastrointestinal disorders) | 15
Abdominal bloating (Gastrointestinal disorders) | 2
Dizziness (General disorders) | 5
Dry eye (Eye disorders) | 4
Dry mouth (Skin and subcutaneous tissue disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 2
Dysphagia (Nervous system disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 10
Edema (Blood and lymphatic system disorders) | 9
Esophagitis (Gastrointestinal disorders) | 1
Gait disturbance (Nervous system disorders) | 3
Fatigue (General disorders) | 14
Neutropenia (Blood and lymphatic system disorders) | 11
Fever (General disorders) | 10
Flushing (Blood and lymphatic system disorders) | 2
Gastrointestinal - other (Gastrointestinal disorders) | 11
Hyperglycemia (Endocrine disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 3
Hemoglobin (Blood and lymphatic system disorders) | 11
Bleeding - other (Blood and lymphatic system disorders) | 3
Hepatobiliary/pancreas - other (Hepatobiliary disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hypertension (General disorders) | 11
Hypotension (General disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Infection (Infections and infestations) | 11
Insomnia (General disorders) | 8
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 16
Lymphatics - other (Blood and lymphatic system disorders) | 2
Hypomagnesemia (Blood and lymphatic system disorders) | 15
Anxiety (Psychiatric disorders) | 10
Depression (Psychiatric disorders) | 3
Mucositis/stomatitis (Skin and subcutaneous tissue disorders) | 14
Metabolic - other (Metabolism and nutrition disorders) | 7
Musculoskeletal - weakness/other (Musculoskeletal and connective tissue disorders) | 3
Sinus reaction (Respiratory, thoracic and mediastinal disorders) | 1
Nausea (Gastrointestinal disorders) | 16
Neurology - other (Nervous system disorders) | 3
Neuropathy (Nervous system disorders) | 2
Neutrophils/Granulocytes (Blood and lymphatic system disorders) | 13
Pain (General disorders) | 16
Kidney perforation (Renal and urinary disorders) | 1
Petichiae/Purpura (Blood and lymphatic system disorders) | 1
Hypophosphatemia (Blood and lymphatic system disorders) | 1
Platelets (Blood and lymphatic system disorders) | 11
Pneumonitis/Pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 3
Prutitis (General disorders) | 5
Psychosis (Psychiatric disorders) | 2
Pulmonary hypertension (Cardiac disorders) | 1
Pulmonary/Upper respiratory - other (Respiratory, thoracic and mediastinal disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 3
Renal failure (Renal and urinary disorders) | 2
Renal/Genitourinary - other (Renal and urinary disorders) | 5
Rigors/chills (General disorders) | 16
Seizure (Nervous system disorders) | 1
Sexual/reproductive function - other (Reproductive system and breast disorders) | 1
Hypernatremia (Blood and lymphatic system disorders) | 1
Hyponatremia (Blood and lymphatic system disorders) | 2
Somnolence/depressed level of consciousness (General disorders) | 1
Atrial fibrillation (Cardiac disorders) | 3
Tachycardia (Cardiac disorders) | 4
Syncope (General disorders) | 1
Dysgeusia (Gastrointestinal disorders) | 1
Tremor (Nervous system disorders) | 2
Dysuria (Renal and urinary disorders) | 1
Urticaria (Renal and urinary disorders) | 4
Vaginal discharge (Reproductive system and breast disorders) | 1
Vascular - other (Vascular disorders) | 4
Ventricular arrhythmia (Cardiac disorders) | 1
Blurred vision (Eye disorders) | 1
Dysarthria (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 11
Weight gain (Metabolism and nutrition disorders) | 2
Weight loss (Metabolism and nutrition disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes